CLINICAL TRIAL: NCT02994290
Title: Evaluation of the Implementation and Effectiveness of a Pilot Quality Improvement Program to Increase HPV Vaccine Uptake: Inpatient Postpartum HPV Immunization (IPP-HPV) Program
Brief Title: Evaluation of the Implementation and Effectiveness of IPP-HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000020062; 1K07CA230234-01 (NIH)
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: HPV Vaccination
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- receive inpatient HPV vaccine (Experimental): We will select a purposive sample of postpartum women into two groups: those who receive inpatient HPV vaccine and those who decline the inpatient dose to interview until we reach thematic saturation which we anticipate to occur with about 8-10 individuals per group. Patients will be selected to include diverse representation in age, race, ethnicity, and parity.
  Interventions: Drug: HPV vaccine; Behavioral: Inpatient Postpartum HPV Immunization Quality Improvement Program
- decline the inpatient dose (Experimental): We will select a purposive sample of postpartum women into two groups: those who receive inpatient HPV vaccine and those who decline the inpatient dose to interview until we reach thematic saturation which we anticipate to occur with about 8-10 individuals per group. Patients will be selected to include diverse representation in age, race, ethnicity, and parity.
  Interventions: Behavioral: Inpatient Postpartum HPV Immunization Quality Improvement Program

INTERVENTIONS:
Drug: HPV vaccine — After the vaccine is administered (or the patient declines the vaccine), a member of the research team (RA) will approach eligible postpartum women and invite them to participate in individual in-depth interviews.
  Arms: receive inpatient HPV vaccine
Behavioral: Inpatient Postpartum HPV Immunization Quality Improvement Program — The program coordinator (PC) will screen electronic medical records of Women's Center patients admitted to the inpatient postpartum service for IPP-HPV eligibility: women ≤ 26 years of age who have not received all 3 doses.
  Nurses and providers in the Women's Center will be encouraged to discuss the HPV vaccine during prenatal care and recommend postpartum immunization to vaccine eligible women.
  All patients will be provided with a Vaccine Information Sheet as is required by law. A postpartum nurse will then administer the HPV vaccine as routine care prior to discharge (unless the patient refuses). A postpartum provider will be available to answer any questions or concerns as needed.

SUMMARY:
The purpose of the proposed pilot study is to assess the implementation of IPP-HPV immunization at Yale New Haven Hospital (YNHH) and to identify potential barriers to and facilitators of this intervention to optimize its feasibility and effectiveness. It is imperative that innovative interventions be developed to achieve comprehensive utilization of this highly effective vaccine to reduce rates of HPV infection, lower rates of cervical and other HPV associated cancers, and address cancer disparities.

DETAILED DESCRIPTION:
Administration of the HPV vaccine during the inpatient postpartum hospital stay has the potential to be an innovative intervention to improve HPV immunization rates. Following onset of pregnancy, the postpartum period becomes the next available opportunity to immunize with the HPV vaccine, which is safe in breastfeeding women. The benefits of such an intervention include a focus on women engaged with the health care system who are often highly motivated to invest in their personal health.

Specific Aims Aim 1: To evaluate receptivity and concerns of postpartum women with receiving the HPV vaccine during the inpatient postpartum admission as part of the Inpatient Postpartum HPV Immunization Quality Improvement Program (IPP-HPV).

Aim 2: To evaluate receptivity and concerns of healthcare providers with inpatient postpartum HPV immunization as part of IPP-HPV and to identify facilitators of and barriers to its implementation.

Aim 3: To assess the uptake and effectiveness of a Pilot Quality Improvement Program to increase HPV vaccine uptake (IPP-HPV) for Yale New Haven Hospital (YNHH) Women's Center and Center for Women's Health and Midwifery (CWHM) postpartum patients ≤ 26 years of age who deliver at YNHH York Street Campus (YSC) or Saint Raphael Campus (SRC).

ELIGIBILITY:
Inclusion Criteria:

* Women participating in the IPP-HPV Quality Improvement Program:
* Postpartum YNHH Women's Center and CWHM patients
* ≤ 26 years at time of delivery who deliver at YNHH YSC or SRC
* Have not already received 3 doses of the HPV vaccine at time of delivery
* Fluent in English or Spanish
* Able and willing to provide consent

AND

* Yale New Haven Hospital (YNHH) Women's Center and Center for Women's Health and Midwifery (CWHM) postpartum patients
* ≤ 26 years of age
* Delivered at YNHH York Street Campus (YSC) or Saint Raphael Campus (SRC) in the first year of the IPP-HPV program or in the one year preceding implementation of the program

OR

* YNHH inpatient postpartum nurses or Women's Center outpatient postpartum nurses or inpatient or outpatient obstetric providers affiliated with the Women's Center or Center for Women's Health and Midwifery
* Able and willing to provide consent

Exclusion Criteria:

-

Ages: 15 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 817 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangini Sheth, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, Women's Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 787 participants and 30 providers
Groups:
- Receive Inpatient HPV Vaccine; Decline the Inpatient Dose: The investigators will select a purposive sample of postpartum women into two groups: those who receive inpatient HPV vaccine and those who decline the inpatient dose to interview until we reach thematic saturation which we anticipate to occur with about 8-10 individuals per group. Patients will be selected to include diverse representation in age, race, ethnicity, and parity.
  HPV vaccine: After the vaccine is administered (or the patient declines the vaccine), a member of the research team (RA) will approach eligible postpartum women and invite them to participate in individual in-depth interviews.
  Inpatient Postpartum HPV Immunization Quality Improvement Program: The program coordinator (PC) will screen electronic medical records of Women's Center patients admitted to the inpatient postpartum service for IPP-HPV eligibility: women ≤ 26 years of age who have not received all 3 doses.
  Nurses and providers in the Women's Center will be encouraged to discuss the HPV vaccine during prenatal care and recommend postpartum immunization to vaccine eligible women.
  All patients will be provided with a Vaccine Information Sheet as is required by law. A postpartum nurse will then administer the HPV vaccine as routine care prior to discharge (unless the patient refuses). A postpartum provider will be available to answer any questions or concerns as needed.
- Providers: Nurses and providers in the Women's Center will be encouraged to discuss the HPV vaccine during prenatal care and recommend postpartum immunization to vaccine eligible women. All patients will be provided with a Vaccine Information Sheet as is required by law. A postpartum nurse will then administer the HPV vaccine as routine care prior to discharge (unless the patient refuses). A postpartum provider will be available to answer any questions or concerns as needed.
Period: Overall Study
Arm/Group | Receive Inpatient HPV Vaccine | Decline the Inpatient Dose | Providers
Started | 491 | 296 | 30
Completed | 491 | 296 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 787 total eligible participants and 30 providers
Groups:
- Receive Inpatient HPV Vaccine; Decline the Inpatient Dose: The investigators will select a purposive sample of postpartum women into two groups: those who receive inpatient HPV vaccine and those who decline the inpatient dose to interview until a thematic saturation is reached. Patients will be selected to include diverse representation in age, race, ethnicity, and parity.
  HPV vaccine: After the vaccine is administered (or the patient declines the vaccine), a member of the research team (RA) will approach eligible postpartum women and invite them to participate in individual in-depth interviews.
  Inpatient Postpartum HPV Immunization Quality Improvement Program: The program coordinator (PC) will screen electronic medical records of Women's Center patients admitted to the inpatient postpartum service for IPP-HPV eligibility: women ≤ 26 years of age who have not received all 3 doses.
  Nurses and providers in the Women's Center will be encouraged to discuss the HPV vaccine during prenatal care and recommend postpartum immunization to vaccine eligible women.
  All patients will be provided with a Vaccine Information Sheet as is required by law. A postpartum nurse will then administer the HPV vaccine as routine care prior to discharge (unless the patient refuses). A postpartum provider will be available to answer any questions or concerns as needed.
- Total: Total of all reporting groups
Arm/Group | Receive Inpatient HPV Vaccine | Decline the Inpatient Dose | Providers | Total
Number analyzed (Participants) | 491 | 296 | 30 | 817
Age, Continuous [Mean (Standard Deviation); unit: years] — mean age in years at delivery Population: this is for patient participants
  years
    number analyzed (Participants) | 491 | 296 | 0 | 787
    (all) | 22.5 (2.7) | 22.5 (2.7) |  | 22.5 (2.7)
Age, Customized [Count of Participants; unit: Participants] — Population: this data was only collected for providers
  Participants
    Providers age: number analyzed (Participants) | 0 | 0 | 30 | 30
    Providers age: <40 | 0 | 0 | 11 | 11
    Providers age: 41-60 | 0 | 0 | 13 | 13
    Providers age: 61+ | 0 | 0 | 5 | 5
    Providers age: Did not report | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — only post-partum women were eligible, data was not collected for providers Population: was not collected for providers
  Participants
    number analyzed (Participants) | 491 | 296 | 0 | 787
    Female | 491 | 296 | 0 | 787
    Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — 787 participants and 30 providers
  Participants
    Race: Black/African American | 99 | 83 | 1 | 183
    Race: White | 42 | 44 | 22 | 108
    Race: Hispanic | 265 | 109 | 1 | 375
    Race: Other | 48 | 31 | 5 | 84
    Race: Unknown | 37 | 29 | 0 | 66
    Race: Asian | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 491 | 296 | 30 | 787
Preferred Language [Count of Participants; unit: Participants] — data was not collected for providers Population: this data was only collected for participants
  Participants
    number analyzed (Participants) | 491 | 296 | 0 | 787
    English | 244 | 190 | 0 | 434
    Spanish | 168 | 47 | 0 | 215
    Other | 46 | 33 | 0 | 79
    Unknown | 33 | 26 | 0 | 59
Providers Job Title [Count of Participants; unit: Participants] — data was only collected for providers Population: this data was only collected for providers
  Participants
    number analyzed (Participants) | 0 | 0 | 30 | 30
    Registered Nurse | 0 | 0 | 14 | 14
    Certified Nurse-Midwife | 0 | 0 | 5 | 5
    Physician | 0 | 0 | 5 | 5
    Physician Assistant | 0 | 0 | 1 | 1
    Advanced Practice Registered Nurse | 0 | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Count of Eligible Patients Agreeing to Receive a Dose of Vaccine
Description: Data gathered via medical charts for which participants agreed to receive a dose and which did not
Time Frame: 12 months
Population: 787 total eligible participants
Measure: Number; unit: participants
Groups:
- Eligible to Receive Inpatient HPV Vaccine: The investigators will select a purposive sample of postpartum women eligible to receive the inpatient HPV vaccine into two groups: those who receive inpatient HPV vaccine and those who decline the inpatient dose. Participants will be interviewed until a thematic saturation is reached (anticipated to occur with about 8-10 individuals per group).
  HPV vaccine: After the vaccine is administered (or the patient declines the vaccine), a member of the research team (RA) will approach eligible postpartum women and invite them to participate in individual in-depth interviews.
  Inpatient Postpartum HPV Immunization Quality Improvement Program: The program coordinator (PC) will screen electronic medical records of Women's Center patients admitted to the inpatient postpartum service for IPP-HPV eligibility: women ≤ 26 years of age who have not received all 3 doses.
  Nurses and providers in the Women's Center will be encouraged to discuss the HPV vaccine during prenatal care and recommend postpartum immunization to vaccine eligible women.
  All patients will be provided with a Vaccine Information Sheet as is required by law. A postpartum nurse will then administer the HPV vaccine as routine care prior to discharge (unless the patient refuses). A postpartum provider will be available to answer any questions or concerns as needed.
Arm/Group | Eligible to Receive Inpatient HPV Vaccine
Number analyzed (Participants) | 787
participants
  Agreed to Receive IPP-HPV | 686
  Did not agree to receive IPP-HPV Dose | 101

2. Primary Outcome: HPV Vaccine Receptivity Thematic Interview
Description: In-person, in-depth interviews will be conducted prior to discharge home from the postpartum hospitalization. If an in-person interview prior to discharge is not possible, an in-person interview will be conducted at the 6-week postpartum visit. Interviews will be conducted using a semi-structured guide with questions based on Consolidated Framework for Implementation Research (CFIR) constructs. Transcripts will be analyzed to determine common themes and priority domains. Standard analytic methods for qualitative data will be employed. A codebook will be developed based on deductive (theory-driven) constructs from the interview guide and applied to a subset of transcripts. This outcome reflects the number of themes derived from thematic interviews.
Time Frame: up to 6 weeks postpartum
Population: a random sub sample of overall participants that completed the thematic interview
Measure: Number; unit: themes
Groups:
- Receive Inpatient HPV Vaccine; Decline the Inpatient Dose: The investigators will select a purposive sample of postpartum women into two groups to interview until thematic saturation is reached: those who receive inpatient HPV vaccine and those who decline the inpatient dose. Patients will be selected to include diverse representation in age, race, ethnicity, and parity.
  HPV vaccine: After the vaccine is administered (or the patient declines the vaccine), a member of the research team (RA) will approach eligible postpartum women and invite them to participate in individual in-depth interviews.
  Inpatient Postpartum HPV Immunization Quality Improvement Program: The program coordinator (PC) will screen electronic medical records of Women's Center patients admitted to the inpatient postpartum service for IPP-HPV eligibility: women ≤ 26 years of age who have not received all 3 doses.
  Nurses and providers in the Women's Center will be encouraged to discuss the HPV vaccine during prenatal care and recommend postpartum immunization to vaccine eligible women.
  All patients will be provided with a Vaccine Information Sheet as is required by law. A postpartum nurse will then administer the HPV vaccine as routine care prior to discharge (unless the patient refuses). A postpartum provider will be available to answer any questions or concerns as needed.
Arm/Group | Receive Inpatient HPV Vaccine | Decline the Inpatient Dose
Number analyzed (Participants) | 18 | 6
themes | 5 | 5

3. Primary Outcome: Barriers to Receiving the HPV Vaccine Thematic Interview
Description: as for outcome 2
Time Frame: up to 6 weeks postpartum
Population: a random sub sample of participants that completed the thematic interview
Measure: Number; unit: themes
Arm/Group | Receive Inpatient HPV Vaccine | Decline the Inpatient Dose
Number analyzed (Participants) | 18 | 6
themes | 5 | 5

4. Secondary Outcome: Number of Participants Who Received or Did Not Receive a Dose of Vaccine
Description: Data gathered via medical charts for which participants received vaccine as inpatient and which did not.
Time Frame: 12 months postpartum
Population: 787 total eligible participants
Measure: Number; unit: participants
Arm/Group | Eligible to Receive Inpatient HPV Vaccine
Number analyzed (Participants) | 787
participants
  Received IPP-HPV Dose | 491
  Did not receive IPP-HPV Dose | 296

5. Secondary Outcome: Receptivity of Healthcare Providers Thematic Interviews
Description: The in-depth individual interviews will be conducted using a semistructured guide based on Consolidated Framework for Implementation Research (CFIR) constructs. Recorded interviews will be transcribed and transcripts analyzed using standard analytic methods for qualitative data as described above. Provider receptivity of IPP-HPV and perceptions of patient acceptance will be categorized by themes. This outcome reflects the number of themes derived from thematic interviews.
Time Frame: up to 12 months
Population: 30 providers
Measure: Number; unit: themes
Arm/Group | Providers
Number analyzed (Participants) | 30
themes | 5

6. Secondary Outcome: Concerns of Healthcare Providers Thematic Interview
Description: as for outcome 5
Time Frame: up to 12 months
Population: 30 providers
Measure: Number; unit: themes
Arm/Group | Providers
Number analyzed (Participants) | 30
themes | 2

7. Other Pre Specified Outcome: Proportion of Patients Who Are Due for Tdap, Influenza or MMR Vaccines and Received Each.
Description: Data gathered via medical charts
Time Frame: 12 months postpartum
Population: data was not collected for this outcome
Groups:
- Eligible to Receive Inpatient HPV Vaccine: We will select a purposive sample of postpartum women into two groups: those who receive inpatient HPV vaccine and those who decline the inpatient dose to interview until we reach thematic saturation which we anticipate to occur with about 8-10 individuals per group. Patients will be selected to include diverse representation in age, race, ethnicity, and parity.
  HPV vaccine: After the vaccine is administered (or the patient declines the vaccine), a member of the research team (RA) will approach eligible postpartum women and invite them to participate in individual in-depth interviews.
  Inpatient Postpartum HPV Immunization Quality Improvement Program: The program coordinator (PC) will screen electronic medical records of Women's Center patients admitted to the inpatient postpartum service for IPP-HPV eligibility: women ≤ 26 years of age who have not received all 3 doses.
  Nurses and providers in the Women's Center will be encouraged to discuss the HPV vaccine during prenatal care and recommend postpartum immunization to vaccine eligible women.
  All patients will be provided with a Vaccine Information Sheet as is required by law. A postpartum nurse will then administer the HPV vaccine as routine care prior to discharge (unless the patient refuses). A postpartum provider will be available to answer any questions or concerns as needed.
Arm/Group | Eligible to Receive Inpatient HPV Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events were not tracked as it was not part of the study protocol
Arm/Group | Eligible to Receive Inpatient HPV Vaccine
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT02994290/Prot_SAP_000.pdf